CLINICAL TRIAL: NCT00003817
Title: A Randomized Phase II Trial of Acupressure and Acustimulation Wrist Bands for the Prevention of Chemotherapy-Induced Nausea and Vomiting
Brief Title: Acupressure and Acustimulation Wrist Bands for the Prevention of Nausea and Vomiting Caused by Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, University of Rochester NCORP Research Base, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000066969; URCC-U3997; NCI-V99-1528
Record Dates: First submitted 1999-11-01; First posted 2004-03-23 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; nausea and vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — dolasetron; Granisetron; Ondansetron; Tropisetron

INTERVENTIONS:
Drug: dolasetron mesylate
Drug: granisetron hydrochloride
Drug: ondansetron
Drug: tropisetron
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Pressure or nerve stimulation applied to an acupuncture point on the inside of the wrist may help control nausea and vomiting during chemotherapy.

PURPOSE: Randomized phase II trial to study the effectiveness of acupressure and acustimulation wrist bands in treating nausea and vomiting in patients undergoing chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of acupressure and acustimulation as adjuncts to standard serotonin antiemetics in reducing acute nausea (day of treatment) and delayed nausea (1-4 days following treatment) associated with cisplatin or doxorubicin based chemotherapy in cancer patients. II. Evaluate the efficacy of acupressure and acustimulation in reducing acute and delayed vomiting and in improving quality of life in cancer patients. III. Investigate the relationship between expectations for the development of chemotherapy-related nausea/vomiting and its actual occurrence in cancer patients.

OUTLINE: This is a randomized study. Patients are stratified according to chemotherapy agent and research site. Patients are randomized to one of three treatment arms. Arm I: Patients receive standard antiemetic therapy with serotonin receptor antagonists. Arm II: Patients receive standard antiemetic therapy with serotonin receptor antagonists and wear an acupressure wrist band (an elastic band equipped with a small plastic button used to apply pressure to a specific point on the wrist) continuously for 5 consecutive days except when necessary to avoid immersion in water. Patients may wear the band on either wrist, including alternating between wrists if desired. Arm III: Patients receive standard antiemetic therapy with serotonin receptor antagonists and wear an acustimulation wrist band (a portable transcutaneous electrical nerve stimulator (TENS) device) continuously for 5 consecutive days except when necessary to avoid immersion in water. Patients may wear the band on either wrist, including alternating between wrists if desired, and may adjust the intensity of stimulation for optimum effectiveness. All patients complete a questionnaire concerning expectations of nausea and other side effects prior to receiving chemotherapy with cisplatin and doxorubicin. Patients in arms II and III complete this measure after the wrist band is in position. All patients complete a questionnaire and a 5 day diary at home concerning nausea and emesis following the first chemotherapy treatment, and then complete a quality of life questionnaire on the fourth day following treatment.

PROJECTED ACCRUAL: A total of 700 patients will be accrued for this study over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of cancer No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No cardiac pacemaker Other: No clinical evidence of current or impending bowel obstruction Able to understand English

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent interferon Chemotherapy: No prior chemotherapy Concurrent cisplatin or doxorubicin based chemotherapy required No multiple day doses of cisplatin, doxorubicin, hexamethylmelamine, dacarbazine, nitrosourea or streptozocin Other concurrent chemotherapy allowed on 1 or multiple days Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: Serotonin receptor antagonist antiemetic (ondansetron, granisetron, tropisetron, or dolasetron mesylate) required

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 1999-10; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Morrow, PhD, MS, Study Chair — James P. Wilmot Cancer Center
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester Cancer Center, Rochester, New York

REFERENCES:
- [Result] Roscoe JA, Morrow GR, Hickok JT, Bushunow P, Pierce HI, Flynn PJ, Kirshner JJ, Moore DF, Atkins JN. The efficacy of acupressure and acustimulation wrist bands for the relief of chemotherapy-induced nausea and vomiting. A University of Rochester Cancer Center Community Clinical Oncology Program multicenter study. J Pain Symptom Manage. 2003 Aug;26(2):731-42. doi: 10.1016/s0885-3924(03)00254-9. PMID 12906958